CLINICAL TRIAL: NCT03546660
Title: Imaging of the Esophagus Using a SECM Capsule
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are currently working and developing our technology to ensure accurate data collection and safety. We will re-open in the future for recruitment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-P000844
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis; Barrett Esophagus
Keywords: EoE; Eosinophilic Esophagitis; Barrett's Esophagus; Capsule; SECM; Tethered Capsule Endomicroscopy
MeSH Terms: conditions — Eosinophilic Esophagitis; Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SECM capsule imaging (Experimental): Participant will swallow the SECM capsule and the imaging of the esophagus will be performed using a SECM optical system
  Interventions: Device: SECM capsule

INTERVENTIONS:
Device: SECM capsule — Participants will swallow a SECM capsule and the SECM imaging will be performed

SUMMARY:
The goal of this validation study is to compare Spectrally Encoded Confocal Microscopy (SECM) Tethered Capsule Endoscopy (TCE) diagnosis of Eosinophilic Esophagitis to that of standard of care endoscopic biopsy.

DETAILED DESCRIPTION:
Eosinophilic esophagitis is an inflammatory condition of the esophagus that occurs in response to certain foods or allergens. Approximately 300,000 people in the US have EoE, the incidence of newly diagnosed EoE is ~30,000/year, and EoE is found in 5-10% of all patients undergoing upper endoscopy. EoE is associated with debilitating symptoms, and is a common cause of dysphagia, strictures, and food impaction; it may even lead to esophageal perforation. Because of the impact of EoE on quality of life as well as the concern that this disease may progress to esophageal fibrosis with unknown long-term risks, experts recommend that EoE be treated until symptoms and eosinophilic infiltrate are resolved. Because the only objective method for diagnosing EoE is histopathologic assessment of multiple upper endoscopic biopsies, the processes of monitoring the esophagus during therapy and the food reintroduction involve a high number of repeat endoscopies. This process is both time consuming and frustrating for patients and their families. Because the endoscopic biopsy requires conscious sedation, it is also costly, exceeding $1000 per procedure. Given the rapid increase in the number of patients with this disease, there is a compelling need for a less invasive and more cost-effective means of identifying eosinophils in the esophagus.

Based on the extensive experience with Optical Coherence Tomography (OCT) and OFDI, the investigators at Tearney laboratory at MGH have developed a spectrally encoded confocal microscopy (SECM) technology that is able to acquire images at significantly higher frame rates than standard confocal microscopy. This SECM capability enables imaging of large portions of the esophagus at 2-µm resolution in realistic procedure times. Furthermore, the investigators at Tearney laboratory have created a tethered capsule SECM device that can be swallowed and used for EoE screening. The investigators at Tearney laboratory lab performed a pilot study using a SECM capsule on 58 subjects (2013-P-000863). The imaging was successful with no adverse or unanticipated events. SECM endoscopy capsule is similar to the approved endoscopy capsule.

A total of sixty (60) subjects will be recruited for this study. The imaging of the esophagus will be obtained. Subjects will not be sedated for the procedure.

The images obtained by the SECM capsule will be compared to the images obtained by the clinical endoscopy and biopsy. SECM imaging will be used for research purposes only and will not be used for diagnosis purposes.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older who are healthy and have no significant health related issues
* Participants 14 years of age of older who are undergoing evaluation for EoE
* Able to give informed consent or assent as per the age of the subject

Exclusion Criteria:

* Inability to swallow pills and capsules
* Esophageal fistula and/or esophageal strictures with a stricture diameter that is smaller than the diameter of the capsule

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of imaging of the Esophagus using a SECM Capsule | 10 minutes (roughly the amount of time it takes to image the esophagus via SECM capsule)
  comparing SECM imaging of the esophagus obtained with a SECM capsule to histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No